CLINICAL TRIAL: NCT04406805
Title: Concentration of Trimethylamine-N-oxide Versus Echocardiographic, Biochemical and Histopathological Parameters of Heart Failure in Patients With Severe Aortic Stenosis: a Prospective, Observatory Trial
Brief Title: TMAO in Patients With Severe Aortic Stenosis
Acronym: TASTE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Sponsor
Other Study IDs: KB/211/2018
Record Dates: First submitted 2020-05-22; First posted 2020-05-28 (Actual); Last update posted 2020-06-05 (Actual); Status verified 2020-03

CONDITIONS: Aortic Stenosis; Heart Failure
Keywords: Aortic Stenosis; Heart Failure; Trimethylamine; TMAO; Bacterial Metabolites
MeSH Terms: conditions — Aortic Valve Stenosis; Heart Failure | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma and urine samples for trimethylamine-N-oxide analysis with a ultra performance liquid chromatograph coupled with a mass spectrometer
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Severe aortic stenosis: Patients will be enrolled among those who will be (i) aged from 18 to 99 years, (ii) admitted to the hospital due to severe aortic stenosis, and (iii) qualified for treatment with either surgical aortic valve replacement or transcatheter aortic valve implantation
  Interventions: Diagnostic Test: Measurement of plasma and urine trimethylamine-N-oxide concentration

INTERVENTIONS:
Diagnostic Test: Measurement of plasma and urine trimethylamine-N-oxide concentration — Information already included in arm/group descriptions.
  Other Names: N-terminal pro-brain natriuretic peptide measurement, echocardiography, biopsy of a myocardium in patients undergoing surgical aortic valve replacement

SUMMARY:
Trimethylamine N-oxide (TMAO) has recently gained increasing scientific interest in the field of cardiovascular disease, including its role in cell protection against osmotic and hydrostatic stress. Aortic stenosis (AS) is the most common valvular heart disease, affecting about 7.6 million people over 75 years of age in North America and Europe alone. We hypothesized that TMAO plays a role in protection of the cardiomyocytes against pressure overload in patients with AS. The primary aim of this study is to assess the correlation between the serum and urine TMAO concentration, and (i) echocardiographic, (ii) biochemical and (iii) histopathological parameters of heart failure in patients with severe AS. The secondary aim of this study is to evaluate a correlation between the baseline TMAO concentrations and the post-treatment clinical status, as well as the post-treatment echocardiographic and biochemical parameters.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent to participate in the study
* Severe aortic stenosis, defined as aortic valve area <1.0 cm2 or aortic valve area index <0.6 cm2/m2 as calculated by the continuity equation on transthoracic echocardiography, regardless of the transvalvular gradient, with or without coexisting symptoms of heart failure
* Qualification for surgical aortic valve replacement or transcatheter aortic valve implantation by the Heart Team in accordance with European Society of Cardiology guidelines

Exclusion Criteria:

* Heart failure of etiology other than aortic stenosis
* Coexisting, haemodynamically significant aortic regurgitation
* Myocardial infarction within the last 3 months
* Coronary revascularization within the last month or planned during transcatheter aortic valve implantation or surgical aortic valve replacement
* Chronic kidney disease with estimated glomerular filtration rate <45 ml/min/1.73 m2
* Acute gastrointestinal disease within the last month
* Active neoplastic disease
* Chronic inflammatory disease
* Autoimmune disease
* Chronic intestinal disease
* Antibiotic therapy within the last 2 months
* Dietary supplements within the last 7 days

Ages: 18 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients will be enrolled among those who will be (i) aged from 18 to 99 years, (ii) admitted to the 1st Chair and Department of Cardiology or Department of Cardiosurgery, Medical University of Warsaw due to severe AS, and (iii) qualified for treatment with either surgical aortic valve replacement or transcatheter aortic valve implantation.
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2019-01-15 (Actual); Primary Completion 2022-02-15 (Estimated); Study Completion 2023-02-15 (Estimated)

PRIMARY OUTCOMES:
Correlation between the serum and urine trimethylamine N-oxide concentration and aortic valve area index | January 15, 2019 - February 15, 2023

SECONDARY OUTCOMES:
Correlation between the serum and urine trimethylamine N-oxide concentration and (i) other echocardiographic, (ii) biochemical and (iii) histopathological parameters of heart failure. | January 15, 2019 - February 15, 2023
Correlation between the baseline trimethylamine N-oxide concentrations and the post-treatment clinical status, as well as the post-treatment echocardiographic and biochemical parameters. | January 15, 2019 - February 15, 2023

CONTACTS AND LOCATIONS:
Locations (1):
- 1st Chair and Department of Cardiology and Department of Cardiosurgery, Medical University of Warsaw, Warsaw, Masovia, Poland

IPD SHARING:
Plan to Share IPD: Undecided
The individual participant shared only in case the identity of the participant has been made unrecognizable.

REFERENCES:
- [Result] Jaworska K, Hering D, Mosieniak G, Bielak-Zmijewska A, Pilz M, Konwerski M, Gasecka A, Kaplon-Cieslicka A, Filipiak K, Sikora E, Holyst R, Ufnal M. TMA, A Forgotten Uremic Toxin, but Not TMAO, Is Involved in Cardiovascular Pathology. Toxins (Basel). 2019 Aug 26;11(9):490. doi: 10.3390/toxins11090490. PMID 31454905